CLINICAL TRIAL: NCT04337008
Title: Renin Angiotensin System - CoronaVirus
Acronym: SRA-COV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-16; 2020-A00795-34 (Other: ANSM)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive COVID 19 patient with no respiratory distress (Active Comparator)
  Interventions: Other: blood draw
- Positive COVID 19 patient with respiratory distress (Experimental)
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — 20 mL blood draw will be performed at J1 et J7

SUMMARY:
The aim of the study is to demonstrate overactivation of Renin Angiotensine System (RAS) in positives COVID-19 patient, especially in those with the most serious clinical forms where the mortality of patients in intensive care is on average 50%.

We are expecting two groups: a group of 25 positive COVID 19 patients in intensive care and a group of 25 positive COVID 19 hospitalized patients in conventional hospitalisation. We will measure RAS, serum potassium and collect data on the treatment of these patients (especially antihypertensive therapy) one week apart (at the patient'entry into hospital and 7 days later).

This is a preliminary study that could possibly allow the start of a therapeutic trial in order to test the effectiveness of RAS blocker treatments in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID 19 patients hospitalized in conventionnal hospitalisation
* Patients hospitalized in intensive care secondary to COVID-19 : Patient under invasive mechanical ventilation (PaO2 / FiO2 ratio <300; PEEP> = 5 cmH20; PCR SARS-CoV-2 positive in a pharyngeal or respiratory sample; PaO2 / FiO2 ratio> 300)

Exclusion Criteria:

* Minor patient
* Patient deprived of liberty
* Patient's refusal to participate in the study
* Patient for whom therapeutic limitation measures such as non-admission to intensive care have been issued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-06-03 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
overactivity of the renin / aldosterone system | 7 days
  demonstrate overactivity of RAS in patients hospitalised in intensive car secondary to COVID-19 compared to control patients (COVID -19 hospitalised patients without complications ).

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido-Pradalie, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX de MARSEILLE
Locations (1):
- ASSISTANCE PUBLIQUE HÖPITAUX de MARSEILLE, Marseille, France

IPD SHARING:
Plan to Share IPD: No